CLINICAL TRIAL: NCT00471588
Title: Dopamine D2/D3 Receptor Agonist and Antagonist Drug Effects on Fronto-striatal Systems Related to Compulsive Behaviour in Healthy Volunteers and Patients With Addictive and Compulsive Disorders
Brief Title: Characterize The Modulatory Effects Of Dopamine D2/D3 Receptor Agonist And Antagonist Drugs On Compulsive Behaviors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: TMT106512
Record Dates: First submitted 2007-05-08; First posted 2007-05-10 (Estimated); Last update posted 2014-09-15 (Estimated); Status verified 2014-09

CONDITIONS: Obsessive-Compulsive Disorder
Keywords: Dopamine; OCD; MRI; stimulant users
MeSH Terms: conditions — Obsessive-Compulsive Disorder | interventions — Pramipexole; Amisulpride

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Pramipexole, Amisulpride — Study Drug
  Other Names: Pramipexole; Amisulpride

SUMMARY:
3 groups of subjects (healthy controls, OCD subjects and stimulant-dependent subjects) will receive pramipexole (1.5 mg, single dose), amisulpride (400 mg, single dose) or placebo in a cross-over, double-blind, placebo-controlled design.

Effects of compulsive behaviour will be assessed using fMRI and cognitive testing.

Assess biomarkers including cardiovascular responses and plasma levels. All groups studied on 3 separate occasions following screening, with at least a week intervening between consecutive assessments. The procedures to be adopted for study assessment will be identical on each occasion.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, between 18 - 55 years of age; the groups will be matched for either handedness.
* Participants must have the ability to comprehend the key components of the consent form and provide informed consent.
* Participants must lead and write (in English) at a level sufficient to complete study related assessments.
* Assessment by a psychiatrist or psychologist, which includes a face-to-face evaluation of the individual using the DSM-VI diagnosis.
* No history of neurological disorder, head/brain injury, hepatitis, or visual impairment.
* No MRI contra-indications (metal in body, claustrophobia) and able to provide blood samples (venous accessibility, especially relevant for drug users).
* Patients with obsessive-compulsive disorder will have a minimum 2-year history of compulsive behaviours satisfying DSM-IV-TR criteria for OCD.
* Participants with chronic stimulant use will have a minimum 2-year history of dependence on class A stimulants, with age of drug abuse onset before 20 years, and will satisfy DSM-IV-TR criteria for dependence on stimulant drugs.
* Control volunteers have to be in good mental and physical health.

Exclusion Criteria:

* A personal history of psychiatric or neurological disorders, as defined by the DSMIV (except OCD in patients with OCD and substance dependence in drug users)
* A history or presence of alcohol / substance abuse or dependence (other than nicotine), as defined by the DSM-IV-TR (except drug dependence group).
* A BDI-II total score greater than 14 will lead to exclusion from the study.
* Treatment with methadone or buprenorphine may interfere with the experimental tasks, and therefore, will lead to exclusion from the study.
* Participants who have any laboratory abnormality that in the investigator's judgement is considered to be clinically significant and could potentially affect subject safety or study outcome.

  * History of clinically significant or current renal dysfunction.
  * Clinically significant abnormalities in hematology, blood chemistry, MRI, urinalysis or physical examination not resolved by baseline visit.
  * Impaired liver function at baseline or history of liver dysfunction.
  * Female participant is pregnant or currently breastfeeding.
* Any serious medical disorder or condition that would in the Investigator's opinion, preclude the administration of study medication and or a history of clinically significant hepatic, cardiac, renal, neurologic, cerebrovascular, metabolic or pulmonary disease.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2006-08; Primary Completion 2007-12 (Actual); Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
Investigate that drug addicts or OCD patients will show similar abnormalities of compulsive behaviour and functional activation of ventral fronto-striatal systems. MRI scans will occur on Wk 1, 2 and 3. Neuropsychological testing Wk 1, 2 and 3. | on Wk 1, 2 and 3

SECONDARY OUTCOMES:
Test the prediction that a dopamine D2/D3 agonist drug (pramipexole)by PK levels. PK sample taken on Week 1 only. | on Week 1 only.
Measure of brain functional activation at rest. | up to week 3
Measure of behavioural performance | up to week 3
Measure of peripheral blood for gene expression and proteomic changes. | up to week 3
Genetic variation in selected genes | up to week 3
Clinical measures (SSRS, SSR, BL-VAS, BDI-II) | up to week 3

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Cambridge, Cambridgeshire, United Kingdom